CLINICAL TRIAL: NCT00524589
Title: Phase II Study of Weekly Intravenous 1,25 Dihydroxycholecelciferol (Calcitriol) + Dexamethasone in Androgen Independent Prostate Cancer
Brief Title: Calcitriol and Dexamethasone in Treating Patients With Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed due to futility
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000563197; RPCI I-65405 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexamethasone and Calcitriol (Experimental): Patients receive oral dexamethasone once on days 1 and 2 and calcitriol IV over 1 hour on day 2. Treatment repeats weekly.
  Interventions: Dietary Supplement: calcitriol; Drug: dexamethasone; Genetic: protein expression analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: calcitriol — IV
Drug: dexamethasone — Oral
Genetic: protein expression analysis — Correlative Study
Other: laboratory biomarker analysis — Correlative Study

SUMMARY:
RATIONALE: Calcitriol may help prostate cancer cells become more like normal cells, and to grow and spread more slowly. Dexamethasone may help calcitriol work better by making tumor cells more sensitive to the drug. Giving calcitriol together with dexamethasone may be an effective treatment for prostate cancer that did not respond to hormone therapy .

PURPOSE: This phase II trial is studying how well giving calcitriol together with dexamethasone works in treating patients with prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the response rate in patients with androgen-independent prostate cancer treated with calcitriol and dexamethasone.
* To evaluate the toxicity of high-dose calcitriol and dexamethasone in these patients.

OUTLINE: Patients receive oral dexamethasone once on days 1 and 2 and calcitriol IV over 1 hour on day 2. Treatment repeats weekly in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and on days 2 and 3 to assess VDR and CYP24 expression in peripheral blood mononuclear cells.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of androgen-independent prostate cancer

  * Evidence of rising PSA level (with or without new lesion by radiograph or physical examination), defined as follows:

    * PSA level > 5 ng/mL and clearly rising on 2 measurements taken ≥ 2 weeks apart after androgen deprivation therapy (i.e., orchiectomy or luteinizing hormone-releasing hormone [LHRH] analogue) and antiandrogen withdrawal, if appropriate
  * PSA rising before and on the first value taken at 4 or 6 weeks after antiandrogen cessation is considered disease progression
* Measurable or evaluable disease as defined by any of the following:

  * Measurable or evaluable tumor masses by radiograph or physical examination
  * Evaluable PSA
* Concurrent LHRH analogue or diethylstilbestrol (DES) for testicular androgen suppression required if no prior bilateral orchiectomy

  * Patients receiving other monotherapy for testicular androgen suppression must switch to a LHRH analogue or DES ≥ 14 days prior to study entry

PATIENT CHARACTERISTICS:

* ECOG 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin > 8.9 g/dL (transfusion or erythropoietin support allowed)
* Serum creatinine ≤ 1.8 mg/dL
* AST ≤ 4 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 mg/dL
* Serum corrected calcium < ULN
* No history of nephrolithiasis within the past 5 years
* No unstable, uncontrolled peptic ulcer disease, congestive heart failure, glaucoma, HIV, or diabetes

PRIOR CONCURRENT THERAPY:

* At least 28 days since prior androgen deprivation therapy (≥ 42 days for bicalutamide)

  * A 28-day washout period is not required for patients who have previously progressed despite antiandrogen withdrawal and who have resumed antiandrogens without reduction of PSA
* At least 14 days since prior radiotherapy
* At least 28 days since prior strontium 89
* At least 28 days since prior chemotherapy and/or investigational agents
* No concurrent medications or supplements that contain additional calcium (e.g., Tums)
* No concurrent radiotherapy for pain control or any other indication
* Concurrent bisphosphonates allowed provided dose/regimen is stable

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone and Calcitriol
Started | 18
Completed | 0
Not Completed | 18
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 16

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Dexamethasone and Calcitriol
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (11.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete or Partial Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: All treated and eligible patients
Measure: Number; unit: percentage of participants
Arm/Group | Dexamethasone and Calcitriol
Number analyzed (Participants) | 18
percentage of participants | 0

2. Secondary Outcome: Corrected Serum Calcium Expression
Description: Number of patients with corrected serum calcium levels between 11 mg/dL and 12 mg/dL detected on 1 or more occasions.
Time Frame: 1 year
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone and Calcitriol
Number analyzed (Participants) | 18
Participants | 6

ADVERSE EVENTS:
Arm/Group | Dexamethasone and Calcitriol
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone and Calcitriol (N=18)
Angina pectoris (Cardiac disorders) | 1 (2)
Arrhythmia (Cardiac disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Chest pain (General disorders) | 1 (2)
Heart rate irregular (Investigations) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone and Calcitriol (N=18)
Anaemia (Blood and lymphatic system disorders) | 8 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4)
Vision blurred (Eye disorders) | 1 (2)
Visual disturbance (Eye disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (8)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 1 (2)
Asthenia (General disorders) | 1 (2)
Chest pain (General disorders) | 2 (4)
Fatigue (General disorders) | 7 (18)
Oedema peripheral (General disorders) | 2 (4)
Pain (General disorders) | 1 (2)
Pyrexia (General disorders) | 2 (4)
Infection (Infections and infestations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Blood albumin decreased (Investigations) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (6)
Blood bilirubin increased (Investigations) | 1 (2)
Blood creatine increased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 4 (18)
Blood urea (Investigations) | 1 (2)
Blood urea increased (Investigations) | 3 (6)
Blood urine present (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 8 (44)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (24)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (10)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4)
Headache (Nervous system disorders) | 1 (2)
Sinus headache (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (4)
Haematuria (Renal and urinary disorders) | 2 (6)
Micturition urgency (Renal and urinary disorders) | 2 (6)
Urinary hesitation (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (2)
Dermabrasion (Surgical and medical procedures) | 1 (2)
Flushing (Vascular disorders) | 4 (9)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes